CLINICAL TRIAL: NCT04140708
Title: Effects of Exercise on Glymphatic Functioning and Neurobehavioral Correlates in Parkinson's Disease
Acronym: FIGHTPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniel Claassen, Associate Professor, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191206; GRANT12719996 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Parkinson's Disease and Parkinsonism; Glymphatic System
Keywords: Exercise; Parkinson's; Glymphatic System
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise--Rock Steady Boxing class (Experimental): Participants will be going twice a week to a Rock Steady Boxing class for an hour/class. Participants will be going to this class for a total of three months.
  Interventions: Behavioral: Exercise--Rock Steady Boxing class

INTERVENTIONS:
Behavioral: Exercise--Rock Steady Boxing class — Rock Steady Boxing is a class designed specifically for those with Parkinsonism and movement difficulty using explosive and fine tuned movements as well as cognitive learning skills.

SUMMARY:
This study is designed to measure the change in patients diagnosed with Parkinson's disease (PD) before, during and after a 12 week exercise program.The focus of this study is the glymphatic system. The glymphatic system is a recentlydiscovered novel waste clearance pathway, in patients with Parkinson's Disease (PD).The glymphatic system acts as a waste-clearance system in the brain of vertebrate animals.The glymphatic system has been proposed in which new clearance pathways involving communication between paravascular spaces, interstitial fluid, and ultimately meningeal and dural lymphatic vessels exists, and we have provided evidence that this system may be dysfunctional in patients with Parkinson's disease with cognitive disorders. Early research suggest glymphatic function increases following exercise, this response is believed to clear beta-amyloid in the brain and may mediate the neurobehavioral response to exercise in PD.

This study will use cognitive exams, neurological exams as well as specialized imaging to record data points and evaluate the glymphatic function after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Participant has Parkinson's disease as defined by the UK Brain Bank Criteria.

  * Patient has demonstrated a positive levodopa or related therapy response.
  * Participant is willing and able to participate in a Rock Steady Boxing class.
  * Participation reports a typically sedentary lifestyle in the 6 months prior to enrollment, i.e., no daily-to-weekly, guided, aerobic or non-aerobic exercise routine.
  * Participant agreeable to an overnight dopaminergic medication washout period.
  * Subject has an identified, reliable method of attending study appointments and Rock Steady Boxing classes.

Exclusion Criteria:

* Clinical Dementia Rating scale score <=1
* Any contraindication or inability to tolerate brain magnetic resonance imaging (MRI) or medical conditions that may interfere with their ability to enter the scanner and/or interfere with interpretation of acquired MRI scanning data (e.g., a pacemaker or any other implanted device or condition that would preclude proximity to a strong magnetic field).
* Any contraindication to overnight dopaminergic medication washout period.
* Any contraindication to participation in Rock Steady Boxing.
* Subject resides at a skilled nursing or dementia care facility, or admission to such a facility is planned during the study period.
* Signs or symptoms of untreated obstructive sleep apnea (i.e., 3+ of the 8 STOP-Bang OSA items). Treatment-compliant OSA patients will not be excluded.
* Signs of MSA, probable Alzheimer disease (according to National Institute of Neurological and Communicative Disorders and Stroke, and the Alzheimer's Disease and Related Disorders), probable vascular dementia (history of cognitive decline concurrent with evidence of cerebrovascular disease progression on neuroimaging).
* Evidence of any clinically significant neurological disorder including but not limited to motor neuron disease or Amyotrophic Lateral Sclerosis (ALS), normal pressure hydrocephalus, brain tumor, seizure disorder, multiple sclerosis, or known structural brain abnormalities.
* History of severe or repeated head injury.
* History of encephalitis.
* Subject has had a significant illness or infection requiring medical intervention in the past 30 days.
* History of neuroleptic use (with the exception of pimivanserin, clozapine or quetiapine) for a prolonged period of time or within the past 6 months.
* Any clinically significant hematological, autoimmune, endocrine, cardiovascular, neoplastic, renal, gastrointestinal, or other disorder that, in the Investigator's opinion, could interfere with the subject's participation in the study, place the subject at increased risk, or confound interpretation of study results.
* Current enrollment in another interventional clinical study involving a therapeutic agent.
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Claassen, MD, Principal Investigator — Associate Professor
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise--Rock Steady Boxing Class
Started | 37
Completed | 28
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.22 (6.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Beta-Amyloid Levels
Description: Using MRI/PET scans to measure change from baseline to followup of beta-amyloid levels
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: SUVr
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 26
SUVr | 0.016675963 (0.037511718)

2. Primary Outcome: Change in Hopkins Verbal Learning Test (HVLT) Scores
Description: HVLT measures verbal learning skills and memory, highest score is 36 and lowest score is 0. The higher score demonstrates better recall/recognition abilities with verbal learning.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 26
score on a scale
  HVLT | 1.67 (3.83)
  HVLT Delayed Recall | 0.78 (1.78)

3. Primary Outcome: Change in Movement Disorder Society--Unified Parkinson's Disease Rating Scale Part III (MDS-UPDRS)
Description: UPDRS measures ease of movement. Highest Score is 108, lowest score is 0. The higher the score, the more difficult movement is for patient.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 26
score on a scale | 2.79 (14.10)

4. Primary Outcome: Mini-Balence Evaluation Systems Test (BESTest)
Description: Mini-BESTest describes movement ability and balance in different scenarios. Highest score is 28, lowest score is 0. The higher the score, the better balance/movement in different conditions.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 26
score on a scale | 4.00 (3.64)

5. Primary Outcome: Freezing of Gait Questionnaire (FOG-Q)
Description: Measures walking gait and how stable it is. Highest score is 24, lowest is 0. The higher the score, the worse walking gait is.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 19
Units on a scale | 0.1052631578947 (0.6578362547106)

6. Primary Outcome: Trail Making Test A&B (TMT)
Description: TMT measures executive functioning and error detection. Measured with time to complete trails. Higher time to complete means more difficulty with executive functioning.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 26
score on a scale
  TMT A | 3.94 (24.99)
  TMT B | 2.82 (50.78)

7. Primary Outcome: Letter Fluency (FAS)
Description: FAS measures how many words a patient can list in a minute beginning with a certain letter (F, A, or S), relating to verbal learning and executive function. The lowest score is 0 words, and the more words listed in a minute beginning with each letter, the better executive functioning. FAS is a unitary neuropsychometric test composed of sub-tasks (F, A, S). The individual scores should not be / are not interpreted.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 26
score on a scale | 1.57 (6.86)

8. Primary Outcome: Simon Task
Description: The Simon task is another well-validated measure of inhibitory action control which has also been studied extensively in PD. This is a conflict task which measures the effect of interfering impulses on the ability to select a goal response. Scores are measured in % accuracy from 0-100, and reaction times from 0 ms and upward per item. The higher the accuracy and lower the reaction time, the better the inhibitory action control and executive functioning.
  The outcome we used is mean and standard deviation of reaction time (seconds) for items correctly responded to.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 18
seconds | 1.2777777777777 (5.3556518310984)

9. Primary Outcome: Patient Recorded Outcomes Measurement Information System-Sleep Disturbance (PROMIS-Sleep)
Description: The PROMIS measures sleep disturbance and impairment. The lowest score is an 8 and the highest is a 40. The higher the score, the worse sleep impairment or disturbance is.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 26
score on a scale
  PROMIS-SRI | -0.21 (5.47)
  PRMIS-SD | -1.18 (5.62)

10. Primary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: The HADS measures anxious and depressive feelings in patients. There are 2 parts, Anxiety, where the lowest score would be a 0 and the highest is 21, and the higher a score is, the more anxious behaviors there are. The second part is a depressive behavior scale, which the lowest score is 0, and the highest is 21, and the higher the score, the more depressive behaviors there are.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 26
score on a scale
  HADS-A | -0.07 (2.58)
  HADS-D | -0.64 (2.44)

11. Primary Outcome: Stroop Interference Task
Description: The stroop interference task measures Measures completion time and number of errors, both corrected and not corrected, and total errors. The low and high scores are patient dependent upon performance, and the higher the scores, the more errors have been made and the worse executive functioning. The amount of time taken on the Stroop task also correlates to having worse executive functioning with a higher completion time.
Time Frame: baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 26
score on a scale
  Stroop-Color | 2.83 (5.91)
  Stroop-Word | 3.68 (13.71)
  Stroop-Color/Word | 3.38 (5.75)

12. Secondary Outcome: ActiGraphy
Description: Measures movement patterns during daily activities and exercise. This is measured in steps taken and movement sensors. The higher amount of steps and activity, the more that they are being active and doing exercise.
Time Frame: continuous between baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: average step count
Arm/Group | Exercise--Rock Steady Boxing Class
Number analyzed (Participants) | 28
average step count | 8314.22 (2904.98)

ADVERSE EVENTS:
Time Frame: 12 weeks per patient participation
Arm/Group | Exercise--Rock Steady Boxing Class
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 2/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise--Rock Steady Boxing Class (N=37)
tracer synthesis issue (Investigations) | 2 (2) — tracer not being synthesized and tested correctly

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT04140708/Prot_001.pdf
  • Statistical Analysis Plan (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT04140708/SAP_002.pdf
  • Informed Consent Form (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT04140708/ICF_000.pdf